CLINICAL TRIAL: NCT02249988
Title: Phase IIB-III Efficacy Study of ABX203 Vaccine as an Adjunct Therapy to Nucleos(t)Ide Analogs to Maintain Control of HBV Replication After Cessation of Treatment in HBeAg Negative Patients With Chronic Hepatitis B
Brief Title: Clinical Efficacy of ABX203 Therapeutic Vaccine in HBeAg Negative Patients With Chronic Hepatitis B
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Abivax S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ABX203-002
Record Dates: First submitted 2014-09-19; First posted 2014-09-26 (Estimated); Last update posted 2017-01-24 (Estimated); Status verified 2015-09

CONDITIONS: Chronic Hepatitis B
MeSH Terms: conditions — Hepatitis B, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1 - ABX203 therapeutic Hepatitis B vaccine treatment arm (Experimental): ABX203 therapeutic vaccine in addition to NUCs background therapy
  Interventions: Drug: ABX203 therapeutic Hepatitis B vaccine treatment arm
- Group 2 - Control arm (No Intervention): NUCs background therapy only

INTERVENTIONS:
Drug: ABX203 therapeutic Hepatitis B vaccine treatment arm
  Arms: Group 1 - ABX203 therapeutic Hepatitis B vaccine treatment arm

SUMMARY:
The study is an open-label, randomized, comparative, multicenter clinical trial. The purpose of this study is to assess the efficacy of ABX203, a new chronic hepatitis B therapeutic vaccine administered as an adjunct therapy to nucleos(t)ide analogs (NUCs), in maintaining control of Hepatitis B disease after cessation of treatment with NUCs in subjects with HBeAg negative chronic Hepatitis B.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subject between 18 and 65 years of age at the time of randomization.
* Must be HBeAg negative and anti-HBe Abs positive for at least 1 year prior to screening and at screening.
* Has HBV DNA < 40 IU/mL for at least 1 year prior to screening and at screening
* Has both ALT and AST levels ≤ ULN for at least 1 year prior to screening and at screening.
* Must be HBsAg positive at screening.
* Has been treated with NUCs for at least 2 years prior to screening.
* Has not been treated with PEG-IFN or IFN for at least 1 year prior to screening.
* For all females, must have a negative serum pregnancy test at screening. For female of childbearing potential, must have been using adequate contraception and must agree to continue to use it during all study period and for 6 months after completion of the study product administration.
* Has provided written informed consent.

Exclusion Criteria:

* Has elevated blood levels of alpha-fetoprotein (AFP) (> 500 ng/mL).
* Has cirrhosis, defined as

  * platelet count < 150,000/mm3, with esophageal varices on imaging and spleen size > 12, or
  * liver stiffness of 11 kilopascal [kPa] as measured by elastography using FibroScan® or .an AST to Platelet Ratio Index (APRI) > 2).
* Has hepatocellular carcinoma (HCC) (diagnosed by ultrasonography).
* Has liver decompensation (albumin < 3.5 g/dL and bilirubin ≥1.3 mg/dL).
* Is Hepatitis C virus (HCV) Ab positive at screening.
* Is Hepatitis delta virus (HDV) Ab positive at screening.
* Is Human Immunodeficiency Virus (HIV) Ab positive at screening.
* Has an immune suppressive disorder or treatment with immunosuppressive drugs.
* Has been treated with corticosteroids within 12 weeks prior to the first administration of study product, with the exception of topical or inhaled corticosteroids.
* Has been treated with rituximab.
* Has other hepatic diseases of different etiology (such as auto-immune hepatitis, toxic hepatitis, Wilson disease, alcoholic or hemochromatosis).
* Has a history of allergic disease or reactions likely to be exacerbated by any component of the study products.
* Has a history of a substance abuse (drug or alcohol) problem within the previous 3 years.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 261 (Actual)
Dates: Start 2014-12; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Percentage of subjects with viral load < 40 IU/mL at Week 48. | Week 48

SECONDARY OUTCOMES:
Clinical response defined as changes in viral load, liver function, time to relapse | Week 48 and Week 96
Immune response defined as T-cell response by ICS (CD4 and CD8 to HBcAg and HBsAg) | Week 48
Safety assessment will be conducted throughout the study and will include physical examinations, vital signs, clinical laboratory évaluations, and the recording of AEs | Participants will be followed for the duration of their study participation up to 96 weeks

CONTACTS AND LOCATIONS:
Locations (12):
- Australia (9):
  - Royal Prince Alfred Hospital, Camperdown
  - Monash Medical Centre Clayton, Clayton
  - St Vincent's Hospital Melbourne, Fitzroy
  - Austin Hospital, Heidelberg
  - Liverpool Hospital, Liverpool
  - The Alfred Hospital, Melbourne
  - Royal Melbourne Hospital, Parkville
  - Royal Perth Hospital, Perth
  - Westmead Hospital, Westmead
- New Zealand (3):
  - Auckland City Hospital, Auckland
  - Waikato Hospital, Hamilton West
  - Wellington Hospital, Wellington

REFERENCES:
- [Derived] Ohlendorf V, Wubbolding M, Honer Zu Siederdissen C, Bremer B, Deterding K, Wedemeyer H, Cornberg M, Maasoumy B. Limited Value of HBV-RNA for Relapse Prediction After Nucleos(t)ide Analogue Withdrawal in HBeAg-negative Hepatitis B Patients. J Viral Hepat. 2025 Apr;32(4):e14026. doi: 10.1111/jvh.14026. Epub 2024 Oct 19. PMID 39425534
- [Derived] Wubbolding M, Lopez Alfonso JC, Lin CY, Binder S, Falk C, Debarry J, Gineste P, Kraft ARM, Chien RN, Maasoumy B, Wedemeyer H, Jeng WJ, Meyer Hermann M, Cornberg M, Honer Zu Siederdissen C. Pilot Study Using Machine Learning to Identify Immune Profiles for the Prediction of Early Virological Relapse After Stopping Nucleos(t)ide Analogues in HBeAg-Negative CHB. Hepatol Commun. 2020 Nov 5;5(1):97-111. doi: 10.1002/hep4.1626. eCollection 2021 Jan. PMID 33437904